CLINICAL TRIAL: NCT06438302
Title: Effects of Nasal Ventilation on Cerebral and Pulmonary Function in Orally Intubated Patients
Acronym: VENTINA
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240271
Record Dates: First submitted 2024-05-21; First posted 2024-05-31 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Hypoxemic Acute Respiratory Failure
Keywords: nasal ventilation; orotracheal intubation; brain activity
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major mechanically ventilated patients intubated orotracheally: The study population will be adult patients with acute respiratory failure who are orally intubated and sedated. These patients should be free of neurological and psychiatric diseases prior to ICU admission. The choice of this particular population is justified by its exposure to mechanical ventilation and continuous sedation, which are recognized risk factors for brain damage.
  Interventions: Device: EEG activity measurement

INTERVENTIONS:
Device: EEG activity measurement — The nasal ventilation device (placed as part of the research) (AIRVO 2; Fisher and Paykel Healthcare, Auckland, New Zealand) will be positioned via nasal cannulas adapted to the patient's anatomy. The FiO2 will be set at 21% and the flow rate will be fixed at 0 L/min at the inclusion visit. The temperature of the humidified nasal oxygenator will be set at 31°C.
  Six 30-minute experimental conditions will be performed successively: 1) 0 L/min flow, FiO2 21%, 2) 30 L/min flow, FiO2 21%, 3) 30 L/min flow, FiO2 100%, 4) 60 L/min flow, FiO2 21%, 5) 60 L/min flow, FiO2 100%, 6) Negative control.
  At the end of each condition, a 10-minute thoracic electrical impedance tomography recording, a 10-minute EEG recording, a 10-minute cerebral NIRS recording and an instantaneous temporal Doppler velocity measurement will be performed. A blood gas (1.5 mL) will also be taken at the end of each condition.
  Other Names: Post-intubation nasal ventilation; Additional blood samples (from care catheter 1.5 mL); Electrical impedance tomography

SUMMARY:
The passage of air through the nasal cavity generates rhythmic oscillations transmitted by the olfactory bulb to the brain, which induces cerebral activation in functional areas and is associated with better cognitive performance compared to oral breathing. Consequently, the abolition of nasal ventilation in patients intubated via the orotracheal route could have deleterious effects on brain activity. Besides the loss of olfaction, the abolition of nasal ventilation could affect brain activity and respiratory control, consequently altering regional pulmonary ventilation.

The hypothesis of the study is that nasal ventilation through the passage of humidified nasal airflow in patients intubated via the orotracheal route would be associated with modulation of cerebral electrical activity and tissue oxygenation and a modification of regional pulmonary ventilation.

DETAILED DESCRIPTION:
The effects of nasal ventilation on cerebral activity will be studied on orally intubated and sedated patients in six experimental conditions. The first condition consists of nociceptive stimulation of the left upper limb as a negative control. In three conditions, the inspired fraction of oxygen (FiO2) will remain at 21% while applying three different rates of humidified nasal air at 0L/min, 30L/min and 60L/min respectively. The last two conditions consist of applying humidified nasal air at 30L/min and 60L/min with a FiO2 of 100%. The primary objective of this study is to evaluate the effects of high-flow humidified nasal air on electroencephalogram activity (root mean square gamma frequency) in sedated, orally intubated patients. The secondary objectives of the study are to evaluate the effects of high-flow humidified nasal air on cerebral perfusion and oxygenation, gas exchange and regional pulmonary ventilation in the same patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Hypoxemic acute respiratory failure
3. Intubation and mechanical ventilation since less than 4 days
4. PaO2/FiO2 ratio less than 200
5. RASS<-4
6. Consent obtained from next of kin
7. Patient with health insurance

Exclusion Criteria:

1. Central nervous system diseases (stroke, MS, epilepsy)
2. Psychiatric illnesses (psychosis, depression) (indicated on patient's medical record)
3. Hemodynamic instability (noradrenalin>2mg/h)
4. Patient on AME
5. Patients under legal protection (guardianship/curators)
6. Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be adult patients with acute respiratory failure who are orally intubated and sedated. These patients should be free of neurological and psychiatric diseases prior to ICU admission. The choice of this particular population is justified by its exposure to mechanical ventilation and continuous sedation, which are recognized risk factors for brain damage.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Study the effects of nasal ventilation on brain electrical activity using electroencephalogram recording (EEG) in sedated orotracheally intubated patients. | At inclusion (day 1) - step 1 to 6
  EEG spectral density spectrum of gamma frequency.

SECONDARY OUTCOMES:
Study the effects of nasal ventilation on cerebral perfusion | At inclusion (day 1) - step 1 to 6
  This outcome will be assessed by the evaluation of the Index of Pulsatility (IP) (IP=(Vs-Vd)/Vm: Vs: Systolic velocity; Vd: Diastolic Velocity; Vm: Mean Velocity)
Study the effects of nasal ventilation on cerebral tissue oxygenation | At inclusion (day 1) - step 1 to 6
  Cerebral tissue oxygenation (% of O2) measured by NIRS (Near Infrared Spectroscopy) electrodes
Study the effects of nasal ventilation on gas exchange | At inclusion (day 1) - step 1 to 6
  Ratio of PaO2 (partial pressure of O2) /FiO2 (inspired oxygen fraction)
Study the effects of nasal ventilation on gas exchange | At inclusion (day 1) - step 1 to 6
  Evaluation of PaCO2 (partial pressure of CO2) (mmHG)
Study the effects of nasal ventilation on regional lung ventilation distribution | At inclusion (day 1) - step 1 to 6
  Evaluation of impedance variation by thoracic electrical impedance tomography.
Study the effects of nasal ventilation on regional lung ventilation distribution | At inclusion (day 1) - step 1 to 6
  Evaluation of ventilation homogeneity by I thoracic electrical impedance tomography.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive Réanimation - Hôpital Pitié -Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, "Commission nationale de l'informatique et des libertés") do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.